CLINICAL TRIAL: NCT07233889
Title: A Prospective Clinical Study Evaluating the Effectiveness and Safety of Enteral Supplementation With Sodium Dihydrogen Phosphate and Disodium Hydrogen Phosphate Granules for Varying Degrees of Hypophosphatemia
Brief Title: Enteral Supplementation With Sodium Dihydrogen Phosphate and Disodium Hydrogen Phosphate Granules for the Treatment of Hypophosphatemia.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wang xiaorong, Internal medicine physician, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ICU202501
Record Dates: First submitted 2025-09-23; First posted 2025-11-18 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Hypophosphatemia
Keywords: Hypophosphatemia; Sodium Dihydrogen Phosphate and Disodium Hydrogen Phosphate Granules
MeSH Terms: conditions — Hypophosphatemia | interventions — sodium phosphate

STUDY DESIGN:
Intervention Model Description: All participants with hypophosphatemia were enrolled in this study and stratified according to the severity of hypophosphatemia: mild hypophosphatemia (0.65-0.80 mmol/L), moderate hypophosphatemia (0.32-0.64 mmol/L), and severe hypophosphatemia (<0.32 mmol/L). All subjects received differentiated phosphorus supplementation strategies: subjects with mild hypophosphatemia were administered 0.306 mmol/(kg·d); subjects with moderate hypophosphatemia received 0.612 mmol/(kg·d); and subjects with severe hypophosphatemia received 0.816 mmol/(kg·d). During the treatment period, venous blood samples were collected from subjects to measure blood phosphorus levels to evaluate the effect of phosphorus supplementation.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mild Hypophosphatemia Group (Experimental): Mild hypophosphatemia is defined as a serum phosphorus level of 0.65-0.80 mmol/L. For subjects with mild hypophosphatemia, the phosphorus supplementation dose is 0.306 mmol/(kg·d) based on the subject's actual body weight. During treatment, venous blood is drawn daily between 5:00 and 6:00 AM to measure serum phosphorus levels and evaluate the effectiveness of supplementation. The investigator determines the severity of hypophosphatemia based on the day's serum phosphorus level and administers the corresponding phosphorus supplementation dose for mild, moderate, or severe cases.
  Interventions: Drug: Sodium Dihydrogen Phosphate and Disodium Hydrogen Phosphate Granules
- Moderate Hypophosphatemia Group (Experimental): Moderate hypophosphatemia is defined as a serum phosphorus level of 0.32-0.64 mmol/L. For subjects with moderate hypophosphatemia, the phosphorus supplementation dose is 0.612 mmol/(kg·d) based on the subject's actual body weight. During treatment, venous blood is drawn daily between 5:00 and 6:00 AM to measure serum phosphorus levels and evaluate the effectiveness of supplementation. The investigator determines the severity of hypophosphatemia based on the day's serum phosphorus level and administers the corresponding phosphorus supplementation dose for mild, moderate, or severe cases.
  Interventions: Drug: Sodium Dihydrogen Phosphate and Disodium Hydrogen Phosphate Granules
- Severe Hypophosphatemia Group (Experimental): Severe hypophosphatemia is defined as a serum phosphate level <0.32 mmol/L. For subjects with severe hypophosphatemia, the phosphorus supplementation dose is 0.816 mmol/(kg·d) based on the subject's actual body weight. During treatment, venous blood is drawn daily between 5:00 and 6:00 AM to measure serum phosphorus levels and evaluate the effectiveness of supplementation. The investigator determines the severity of hypophosphatemia based on the day's serum phosphorus level and administers the corresponding phosphorus supplementation dose for mild, moderate, or severe cases.
  Interventions: Drug: Sodium Dihydrogen Phosphate and Disodium Hydrogen Phosphate Granules

INTERVENTIONS:
Drug: Sodium Dihydrogen Phosphate and Disodium Hydrogen Phosphate Granules — After signing the informed consent form (ICF), eligible subjects were stratified based on the severity of hypophosphatemia during the screening period: mild hypophosphatemia (0.65-0.80 mmol/L), moderate hypophosphatemia (0.32-0.64 mmol/L), or severe hypophosphatemia (<0.32 mmol/L).
  Following enrollment, subjects entered a treatment period of up to 14 days. All subjects received a differentiated phosphate supplementation strategy based on actual body weight: subjects with mild hypophosphatemia received 0.306 mmol/(kg·d); those with moderate hypophosphatemia received 0.612 mmol/(kg·d); and those with severe hypophosphatemia received 0.816 mmol/(kg·d). During the treatment period, venous blood was drawn daily between 5:00 and 6:00 AM to measure serum phosphorus levels and evaluate the efficacy of supplementation. Based on the daily serum phosphorus level, the investigator determined the severity of hypophosphatemia and administered the corresponding phosphate dose.

SUMMARY:
The purpose of this clinical trial is to evaluate the efficacy and safety of Sodium Dihydrogen Phosphate and Disodium Hydrogen Phosphate Granules for the treatment of participants with mild, moderate, and severe hypophosphatemia. The main questions it aims to answer are:

Does enteral supplementation of Sodium Dihydrogen Phosphate and Disodium Hydrogen Phosphate Granules elevate participants' serum phosphorus? Does enteral supplementation of Sodium Dihydrogen Phosphate and Disodium Hydrogen Phosphate Granules cause gastrointestinal complications? Participants with hypophosphatemia will receive Sodium Dihydrogen Phosphate and Disodium Hydrogen Phosphate Granules orally or via nasogastric tube to observe the efficacy and safety of enteral phosphate supplementation.

Participants will take Sodium Dihydrogen Phosphate and Disodium Hydrogen Phosphate Granules daily, with varying doses based on the severity of hypophosphatemia, for a maximum of 14 days. The effect of phosphate supplementation will be assessed daily through blood draws, and their gastrointestinal symptoms will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-80 years (inclusive), regardless of gender;
2. ICU inpatients with a serum phosphate concentration <0.80 mmol/L, and for whom the clinician determines phosphate supplementation is required;
3. Ability to receive enteral nutrition, with a daily enteral caloric intake ≥10 kcal/kg/day;
4. The subject or their legal guardian fully understands the purpose and significance of this trial, voluntarily agrees to participate, provides written informed consent, and is willing to strictly adhere to the clinical study protocol and complete the study.

Exclusion Criteria:

1. Pregnant and lactating women;
2. Patients with contraindications for enteral administration, such as acute upper gastrointestinal bleeding, mechanical intestinal obstruction, severe acute pancreatitis, digestive tract fistula, gastrointestinal dysfunction, intra-abdominal hypertension, enteral feeding intolerance, or continuous gastrointestinal decompression;
3. Expected ICU stay ≤96 hours;
4. Known allergy to any component of the investigational drug or drugs with a similar chemical structure;
5. Severe renal impairment: estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m²;
6. Subjects with hyperthyroidism requiring clinical intervention;
7. Subjects requiring sodium restriction;
8. Other conditions deemed by the investigator as unsuitable for inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The rate of achieving target serum phosphorus levels (≥0.80 mmol/L) with enteral phosphorus supplementation in patients during the study period. | Within 14 days of study enrollment
  Among patients receiving enteral phosphate supplementation during the study period, the proportion achieving the target serum phosphate level (≥0.80 mmol/L). This proportion ranges from 0% to 100%, with a higher value indicating better treatment efficacy of enteral phosphate supplementation.

SECONDARY OUTCOMES:
The magnitude of serum phosphorus elevation per 1 mmol of enteral phosphorus supplementation in patients during the study period. | The total duration from the start of enteral phosphorus supplementation to the end of phosphorus therapy is less than 14 days.
  The magnitude of serum phosphorus elevation per 1 mmol of enteral phosphorus supplementation in patients during the study period. A greater magnitude of serum phosphorus elevation indicates better treatment efficacy of phosphorus supplementation.
Average time to achieve target serum phosphorus concentration during phosphorus replacement therapy | The total duration from the initiation of enteral phosphate supplementation to the normalization of serum phosphate levels is less than 14 days.
  Average time to achieve target serum phosphorus concentration during phosphorus replacement therapy. A shorter time indicates better efficacy of phosphorus supplementation.
The proportion of patients with a blood phosphorus concentration increase of less than 0.1 mmol/L over any 72-hour period during phosphorus supplementation therapy. | From the initiation of enteral phosphate supplementation to the end of treatment, the increase in serum phosphate levels within any 72-hour period occurs over a total duration of less than 14 days.
  The proportion of patients with a blood phosphorus concentration increase of less than 0.1 mmol/L over any 72-hour period during phosphorus supplementation therapy. This proportion reflects the efficacy of phosphorus replacement therapy, with a higher proportion indicating poorer treatment response in more patients.
Proportion of withdrawals due to intolerance to enteral phosphorus supplementation | During the study period, the maximum duration shall not exceed 14 days.
  Proportion of withdrawals due to intolerance to enteral phosphorus supplementation. A lower withdrawal rate indicates the successful selection of the study population.
Incidence of Adverse Reactions | The entire duration of the study, from initiation to completion, shall not exceed 14 days.
  The incidence of adverse reactions primarily includes discomfort symptoms such as diarrhea, abdominal pain, nausea, and vomiting.
Changes in APACHE II and SOFA scores from baseline | APACHE II and SOFA scores within 24 hours before the start of the study and within 24 hours before the end of the study
  Changes from baseline in the Acute Physiology and Chronic Health Evaluation (APACHE II) score and Sequential Organ Failure Assessment (SOFA) score. The APACHE II score ranges from 0 to 71 points, with higher scores indicating greater mortality risk. The SOFA score ranges from 0 to 24 points, where higher scores reflect more severe organ dysfunction and indicate a more critical patient condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Cheng YC, Beh JY, Wu PH, Tsai NY, Jao SW. Early botulinum toxin injection reduces pain after hemorrhoidectomy: a pilot study. Tech Coloproctol. 2022 Jan;26(1):53-60. doi: 10.1007/s10151-021-02542-4. Epub 2021 Oct 27. PMID 34705137
- [Result] Kaya U, Dal Yilmaz U. Ideal Suggestions for Discharge Training and Telephone Counseling of Patients With Coronary Artery Bypass Graft Surgery: A Randomized Controlled and Experimental Study. J Korean Med Sci. 2022 Sep 5;37(35):e269. doi: 10.3346/jkms.2022.37.e269. PMID 36065653
- [Result] Felsenfeld AJ, Levine BS. Approach to treatment of hypophosphatemia. Am J Kidney Dis. 2012 Oct;60(4):655-61. doi: 10.1053/j.ajkd.2012.03.024. Epub 2012 Aug 3. PMID 22863286
- [Result] Geerse DA, Bindels AJ, Kuiper MA, Roos AN, Spronk PE, Schultz MJ. Treatment of hypophosphatemia in the intensive care unit: a review. Crit Care. 2010;14(4):R147. doi: 10.1186/cc9215. Epub 2010 Aug 3. PMID 20682049
- [Result] Nguyen CD, Panganiban HP, Fazio T, Karahalios A, Ankravs MJ, MacIsaac CM, Rechnitzer T, Arno L, Tran-Duy A, McAlister S, Ali Abdelhamid Y, Deane AM. A Randomized Noninferiority Trial to Compare Enteral to Parenteral Phosphate Replacement on Biochemistry, Waste, and Environmental Impact and Healthcare Cost in Critically Ill Patients With Mild to Moderate Hypophosphatemia. Crit Care Med. 2024 Jul 1;52(7):1054-1064. doi: 10.1097/CCM.0000000000006255. Epub 2024 Mar 25. PMID 38537225
- [Result] Engwerda E, van den Berg M, Blans M, Bech A, de Boer H. Efficacy and safety of a phosphate replacement strategy for severe hypophosphatemia in the ICU. Neth J Med. 2018 Dec;76(10):437-441. PMID 30569887
- [Result] Lair CS, Brown LS, Edwards A, Jacob T, Brion LP, Jaleel M. Quality improvement project in a neonatal intensive care unit reduced the prevalence and duration of hypophosphatemia with significant and sustainable results. Nutr Clin Pract. 2023 Dec;38(6):1379-1391. doi: 10.1002/ncp.10986. Epub 2023 Apr 12. PMID 37042685
- [Result] Rubio-Aliaga I, Krapf R. Phosphate intake, hyperphosphatemia, and kidney function. Pflugers Arch. 2022 Aug;474(8):935-947. doi: 10.1007/s00424-022-02691-x. Epub 2022 May 5. PMID 35511366
- [Result] Dickerson RN, Gervasio JM, Sherman JJ, Kudsk KA, Hickerson WL, Brown RO. A comparison of renal phosphorus regulation in thermally injured and multiple trauma patients receiving specialized nutrition support. JPEN J Parenter Enteral Nutr. 2001 May-Jun;25(3):152-9. doi: 10.1177/0148607101025003152. PMID 11334065
- [Result] Daily WH, Tonnesen AS, Allen SJ. Hypophosphatemia--incidence, etiology, and prevention in the trauma patient. Crit Care Med. 1990 Nov;18(11):1210-4. doi: 10.1097/00003246-199011000-00004. PMID 2225887
- [Result] Cohen J, Kogan A, Sahar G, Lev S, Vidne B, Singer P. Hypophosphatemia following open heart surgery: incidence and consequences. Eur J Cardiothorac Surg. 2004 Aug;26(2):306-10. doi: 10.1016/j.ejcts.2004.03.004. PMID 15296888
- [Result] Hoffmann M, Zemlin AE, Meyer WP, Erasmus RT. Hypophosphataemia at a large academic hospital in South Africa. J Clin Pathol. 2008 Oct;61(10):1104-7. doi: 10.1136/jcp.2007.054940. PMID 18820097